CLINICAL TRIAL: NCT01014481
Title: Initiation of a Once Daily Regimen of Tenofovir, Lamivudine and Efavirenz After 4 Weeks Versus 12 Weeks of Tuberculosis Treatment in HIV-1 Infected Patients (Time Study)
Brief Title: Appropriate Timing of HAART in Co-infected HIV/TB Patients
Acronym: TIME
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: this study was ended prematurely by ethical committees with a reason of the final outcome was achieved with no longer recruitment was needed.
Sponsor: Bamrasnaradura Infectious Diseases Institute (Other Government)
Collaborators: Mahidol University (Other); Thai Red Cross AIDS Research Centre (Other)
Responsible Party: Weerawat Manosuthi, Bamrasnaradura Infectious Diseases Institute, Ministry of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0435.3/1551
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: HIV Infections; Tuberculosis
Keywords: HIV; tuberculosis; antiretroviral treatment; timing
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Tenofovir; Lamivudine; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- start antiretroviral treatment (Experimental): the optimal timing to initiate antiretroviral therapy in HIV-infected patients who are receiving tuberculosis treatment between at 4 weeks and at 12 weeks after tuberculosis treatment
  Interventions: Drug: tenofovir, lamivudine, efavirenz

INTERVENTIONS:
Drug: tenofovir, lamivudine, efavirenz — initiate tenofovir 300 mg/day, lamivudine 300 mg/day, efavirenz 600 mg/day between at 4 weeks and at 12 weeks after tuberculosis treatment
  Other Names: at 4 weeks versus at 12 weeks after tuberculosis treatment

SUMMARY:
To study the optimal timing to initiate antiretroviral therapy in HIV-infected patients who are receiving tuberculosis treatment between at 4 weeks and at 12 weeks after tuberculosis treatment by comparing the composite end point of death rate, hospitalization rate and adverse drug reactions at week 48, 96 and 144.

DETAILED DESCRIPTION:
The growing epidemic of HIV poses a serious public health threat in many countries, including Thailand. Mortality is clearly reduced in HIV and tuberculosis (TB) co-infected patients who initiate antiretroviral therapy (ART) after the treatment of TB, but the optimal timing to initiate ART is one of the major concern for patients concurrently receiving both therapies. To date, the prospective, randomized, control trial to study the optimal timing to initiate ART in the patients is still limited. In addition, the current recommendation to start ART in patients co-infected with HIV and TB is still based on expert opinions. Here, the investigators plan to investigate the optimal timing to initiate antiretroviral therapy in HIV-infected patients who are receiving tuberculosis treatment between at 4 weeks and at 12 weeks after tuberculosis treatment by comparing the composite end point of death rate, hospitalization rate and adverse drug reactions at week 48, 96 and 144 at Bamrasnaradura Infectious Diseases Institute, Ministry of Public Health, Nonthaburi, Thailand.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age
2. HIV-1 infected patients
3. Naïve to antiretroviral treatment
4. Baseline CD4 cell count <350 cells/mm3 at enrolment
5. Diagnosed as having active tuberculosis by clinical features or positive acid fast stain or positive TB culture; and receiving rifampicin containing antituberculous regimen
6. Signed inform consent

Exclusion Criteria:

1. Serum transaminase enzymes ≥ 5 times of upper normal limit or total bilirubin ≥ 3 times of upper normal limit
2. Serum creatinine ≥ 2 times of upper normal limit
3. Lactation or pregnancy
4. Receiving any immunosuppressive agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2009-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
death rate | 48 weeeks

SECONDARY OUTCOMES:
hospitalization | 48 weeks
adverse events | 48 weeks
composite endpoint of a. death b. hospitalization and c. adverse event | 48 weeks
TB IRIS | 48 weeks
Risk of death | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Weerawat Manosuthi, MD, Principal Investigator — Bamrasnaradura Infectious Diseases Institute, Ministry of Public Health, Nonthaburi, Thailand
Locations (1):
- Bamrasnaradura Infectious Diseases Institute, Ministry of Public Health, Nonthaburi, Changwat Nonthaburi, Thailand

REFERENCES:
- [Derived] Kiertiburanakul S, Manosuthi W, Sungkanuparph S. Optimal timing of antiretroviral therapy initiation in patients coinfected with HIV and tuberculosis. Expert Rev Clin Pharmacol. 2011 Mar;4(2):143-6. doi: 10.1586/ecp.11.2. No abstract available. PMID 22115397